CLINICAL TRIAL: NCT05917288
Title: A Multi-Centre, Open-Label Study to Evaluate the Pharmacokinetics and Safety of Subcutaneously Administered Belimumab Plus Standard Therapy in Chinese Pediatric Participants With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of Belimumab in Chinese Pediatric Participants With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 217091
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Belimumab; Pediatric; Pharmacokinetics; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab; Standard of Care

STUDY DESIGN:
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving belimumab + Standard of care (SOC) (Experimental): Participants will receive belimumab 200 milligrams SC injection according the Baseline body weight plus SOC.
  Interventions: Biological: Belimumab; Drug: Standard of care

INTERVENTIONS:
Biological: Belimumab — Belimumab will be administered
Drug: Standard of care — Standard of care will be administered

SUMMARY:
This study will evaluate the pharmacokinetic characteristics and safety of belimumab subcutaneous (SC) in Chinese pediatric participants with SLE who have completed 48 weeks belimumab Intravenous (IV) treatment in 213560 study (NCT04908865)

ELIGIBILITY:
Inclusion Criteria:

* Participants between 5 and 17 years of age inclusive, at the time of informed consent
* Chinese pediatric participants with SLE, who have completed 48 weeks treatment in study 213560 and who, in the opinion of the investigator, may benefit from treatment with GSK1550188.
* Body weight greater than equal to >=15 kilograms (kg), at the time of signing the informed consent.
* Male and/or female:

  1. No contraceptive measures are required for male participants.
  2. Female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

  i) Is a woman of non-childbearing potential OR ii) Is a woman of childbearing potential and using a contraceptive method that is highly effective, with a failure rate of <1%
* Participant signs and dates a written age-appropriate assent form (in accordance with applicable regulations) and the parent or legal guardian (or emancipated minor) that has the ability to understand the requirements of the study, provides written informed consent (including consent for the use and disclosure of research-related health information) that the participant will comply with the study protocol procedures (including required study visits).

Exclusion Criteria:

* Participants who have developed clinical evidence of significant, unstable or uncontrolled, acute or chronic diseases not due to SLE (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious diseases), or experienced an Adverse events (AE) in 213560 study that could, in the opinion of the principal investigator, put the participant at undue risk.
* Have developed any other medical diseases (e.g., cardiopulmonary), laboratory abnormalities, or conditions that, in the opinion of the principal investigator, makes the participant unsuitable for the study.
* Have an estimated glomerular filtration rate as calculated by Schwartz Formula of less than 30 milliliter per minute (mL/min).
* Have an Immunoglobulin A (IgA) deficiency (IgA level <10 milli gram per deciliter [mg/dL]).
* Have a Grade 3 or greater laboratory abnormality based on the protocol toxicity scale except for the following that are allowed:

  1. Stable Grade 3 hypoalbuminemia due to lupus nephritis and not related to liver disease or malnutrition.
  2. Any grade proteinuria
  3. Stable Grade 3 gamma glutamyl transferase (GGT) elevation due to lupus hepatitis and not related to alcoholic liver disease, uncontrolled diabetes or viral hepatitis. If present, any abnormalities in the alanine transaminase (ALT) and/or aspartate aminotransferase (AST) must be <= Grade 2.
  4. Stable Grade 3 neutropenia; or stable Grade 3 lymphopenia; or stable Grade 3 leukopenia, due to SLE.
* Developing a positive test for Human immunodeficiency virus (HIV) antibody after inclusion into 213560, per investigator's discretion according to clinical need.
* Developing hepatitis B: Serologic evidence of Hepatitis B (HB) infection defined as Hepatitis B surface antigen positive (HBsAg+) OR Hepatitis B core antibody positive (HBcAb+) after inclusion into 213560, per investigator's discretion according to clinical need.
* Developing a positive test for Hepatitis C antibody after inclusion into 213560, per investigator's discretion according to clinical need.
* Have received a live or live-attenuated vaccine within 30 Days of Day 1.
* Are unable or unlikely, in the opinion of the investigator, to administer belimumab by SC injection and have no reliable source to administer the injection.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GSK Clinical Trials
Locations (6):
- China (6):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Suzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 16 participants were enrolled in this study.
Pre-assignment Details: Participants who had completed 48 weeks of intravenous (IV) belimumab treatment in study 213560 (NCT04908865) were enrolled in this study.
Groups:
- Belimumab 200 mg/mL: Participants with systemic lupus erythematosus (SLE), who had completed 48 weeks of IV belimumab treatment in study 213560 (NCT04908865), received belimumab 200 milligrams per milliliter (mg/mL) as a subcutaneous (SC) injection over 12 weeks along with standard of care (SOC) therapy. The dosing frequency of belimumab was based on the body weight of the participants. Participants weighing greater than or equal to (>=) 50 kilograms (kg) received belimumab every week, participants weighing between 30 kg and less than (<) 50 kg received belimumab every 10 days, and participants weighing between 15 kg and < 30 kg received belimumab every 2 weeks.
Period: Overall Study
Arm/Group | Belimumab 200 mg/mL
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Belimumab 200 mg/mL: Participants with SLE, who had completed 48 weeks of IV belimumab treatment in study 213560 (NCT04908865), received belimumab 200 mg/mL as an SC injection over 12 weeks along with SOC therapy. The dosing frequency of belimumab was based on the body weight of the participants. Participants weighing >= 50 kg received belimumab every week, participants weighing between 30 kg and < 50 kg received belimumab every 10 days, and participants weighing between 15 kg and < 30 kg received belimumab every 2 weeks.
Arm/Group | Belimumab 200 mg/mL
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 12.9 (2.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve at Steady-state to the End of the Dosing Period (AUCss,0-tau) of Belimumab for Participants Weighing Greater Than or Equal to (>=) 50 Kilograms (kg)
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of belimumab. AUCss,0-tau of belimumab for participants weighing >= 50 kg has been reported. As the first dose of belimumab was administered on Day 1, Week 12 post-dose correlates to Day 1 plus 84 days, i.e., Day 85.
Time Frame: Pre-dose on Days 1, 8, and 78, and post-dose on Days 4, 81, and 85
Population: PK Analysis Set included all participants assigned treatment who received at least one dose of study treatment and for whom at least one post belimumab treatment PK sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*micrograms per milliliter
Groups:
- Belimumab 200 mg/mL Every Week: Participants with SLE, who had completed 48 weeks of IV belimumab treatment in study 213560 (NCT04908865) and weighed >= 50 kg, received belimumab 200 mg/mL as an SC injection every week over 12 weeks along with SOC therapy.
Arm/Group | Belimumab 200 mg/mL Every Week
Number analyzed (Participants) | 10
Days*micrograms per milliliter | 633.26 (27.50)

2. Primary Outcome: Area Under the Curve at Steady-state to the End of the Dosing Period (AUCss,0-tau) of Belimumab for Participants Weighing Between 30 kg and Less Than (<) 50 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. AUCss,0-tau of belimumab for participants weighing between 30 kg and < 50 kg has been reported.
Time Frame: Pre-dose on Days 1, 11, and 71, and post-dose on Days 4, 74, and 81
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*micrograms per milliliter
Groups:
- Belimumab 200 mg/mL Every 10 Days: Participants with SLE, who had completed 48 weeks of IV belimumab treatment in study 213560 (NCT04908865) and weighed between 30 kg and < 50 kg, received belimumab 200 mg/mL as an SC injection every 10 days over 12 weeks along with SOC therapy.
Arm/Group | Belimumab 200 mg/mL Every 10 Days
Number analyzed (Participants) | 5
Days*micrograms per milliliter | 807.57 (17.44)

3. Primary Outcome: Area Under the Curve at Steady-state to the End of the Dosing Period (AUCss,0-tau) of Belimumab for Participants Weighing Between 15 kg and < 30 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. AUCss,0-tau of belimumab for participants weighing between 15 kg and < 30 kg has been reported. As the first dose of belimumab was administered on Day 1, Week 12 post-dose correlates to Day 1 plus 84 days, i.e., Day 85.
Time Frame: Pre-dose on Days 1, 15, and 71, and post-dose on Days 4, 74, and 85
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*micrograms per milliliter
Groups:
- Belimumab 200 mg/mL Every 2 Weeks: Participants with SLE, who had completed 48 weeks of IV belimumab treatment in study 213560 (NCT04908865) and weighed between 15 kg and < 30 kg, received belimumab 200 mg/mL as an SC injection every 2 weeks over 12 weeks along with SOC therapy.
Arm/Group | Belimumab 200 mg/mL Every 2 Weeks
Number analyzed (Participants) | 1
Days*micrograms per milliliter | 1365.23 (NA) — 'NA' indicates that geometric coefficient of variation could not be calculated as only 1 participant was analyzed.

4. Primary Outcome: Average Serum Concentration at Steady State (Cavg,ss) of Belimumab for Participants Weighing >= 50 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. Cavg,ss of belimumab for participants weighing >= 50 kg has been reported. As the first dose of belimumab was administered on Day 1, Week 12 post-dose correlates to Day 1 plus 84 days, i.e., Day 85.
Time Frame: Pre-dose on Days 1, 8, and 78, and post-dose on Days 4, 81, and 85
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 200 mg/mL Every Week
Number analyzed (Participants) | 10
Micrograms per milliliter | 90.47 (27.50)

5. Primary Outcome: Average Serum Concentration at Steady State (Cavg,ss) of Belimumab for Participants Weighing Between 30 kg and < 50 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. Cavg,ss of belimumab for participants weighing between 30 kg and < 50 kg has been reported.
Time Frame: Pre-dose on Days 1, 11, and 71, and post-dose on Days 4, 74, and 81
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 200 mg/mL Every 10 Days
Number analyzed (Participants) | 5
Micrograms per milliliter | 80.76 (17.44)

6. Primary Outcome: Average Serum Concentration at Steady State (Cavg,ss) of Belimumab for Participants Weighing Between 15 kg and < 30 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. Cavg,ss of belimumab for participants weighing between 15 kg and < 30 kg has been reported. As the first dose of belimumab was administered on Day 1, Week 12 post-dose correlates to Day 1 plus 84 days, i.e., Day 85.
Time Frame: Pre-dose on Days 1, 15, and 71, and post-dose on Days 4, 74, and 85
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 200 mg/mL Every 2 Weeks
Number analyzed (Participants) | 1
Micrograms per milliliter | 97.52 (NA) — 'NA' indicates that geometric coefficient of variation could not be calculated as only 1 participant was analyzed.

7. Primary Outcome: Minimum Serum Concentration at Steady State (Cmin,ss) of Belimumab for Participants Weighing >= 50 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. Cmin,ss of belimumab for participants weighing >= 50 kg has been reported. As the first dose of belimumab was administered on Day 1, Week 12 post-dose correlates to Day 1 plus 84 days, i.e., Day 85.
Time Frame: Pre-dose on Days 1, 8, and 78, and post-dose on Days 4, 81, and 85
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 200 mg/mL Every Week
Number analyzed (Participants) | 10
Micrograms per milliliter | 82.63 (28.69)

8. Primary Outcome: Minimum Serum Concentration at Steady State (Cmin,ss) of Belimumab for Participants Weighing Between 30 kg and < 50 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. Cmin,ss of belimumab for participants weighing 30 kg and < 50 kg has been reported.
Time Frame: Pre-dose on Days 1, 11, and 71, and post-dose on Days 4, 74, and 81
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 200 mg/mL Every 10 Days
Number analyzed (Participants) | 5
Micrograms per milliliter | 70.71 (20.14)

9. Primary Outcome: Minimum Serum Concentration at Steady State (Cmin,ss) of Belimumab for Participants Weighing Between 15 kg and < 30 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. Cmin,ss of belimumab for participants weighing 15 kg and < 30 kg has been reported. As the first dose of belimumab was administered on Day 1, Week 12 post-dose correlates to Day 1 plus 84 days, i.e., Day 85.
Time Frame: Pre-dose on Days 1, 15, and 71, and post-dose on Days 4, 74, and 85
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 200 mg/mL Every 2 Weeks
Number analyzed (Participants) | 1
Micrograms per milliliter | 80.95 (NA) — 'NA' indicates that geometric coefficient of variation could not be calculated as only 1 participant was analyzed.

10. Primary Outcome: Maximum Serum Concentration During the Dosing Interval at Steady State (Cmax,ss) of Belimumab for Participants Weighing >= 50 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. Cmax,ss of belimumab for participants weighing >= 50 kg has been reported. As the first dose of belimumab was administered on Day 1, Week 12 post-dose correlates to Day 1 plus 84 days, i.e., Day 85.
Time Frame: Pre-dose on Days 1, 8, and 78, and post-dose on Days 4, 81, and 85
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 200 mg/mL Every Week
Number analyzed (Participants) | 10
Micrograms per milliliter | 93.36 (25.80)

11. Primary Outcome: Maximum Serum Concentration During the Dosing Interval at Steady State (Cmax,ss) of Belimumab for Participants Weighing Between 30 kg and < 50 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. Cmax,ss of belimumab for participants weighing between 30 kg and < 50 kg has been reported.
Time Frame: Pre-dose on Days 1, 11, and 71, and post-dose on Days 4, 74, and 81
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 200 mg/mL Every 10 Days
Number analyzed (Participants) | 5
Micrograms per milliliter | 87.15 (15.91)

12. Primary Outcome: Maximum Serum Concentration During the Dosing Interval at Steady State (Cmax,ss) of Belimumab for Participants Weighing Between 15 kg and < 30 kg
Description: Blood samples were collected at indicated time points for PK analysis of belimumab. Cmax,ss of belimumab for participants weighing between 15 kg and < 30 kg has been reported. As the first dose of belimumab was administered on Day 1, Week 12 post-dose correlates to Day 1 plus 84 days, i.e., Day 85.
Time Frame: Pre-dose on Days 1, 15, and 71, and post-dose on Days 4, 74, and 85
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 200 mg/mL Every 2 Weeks
Number analyzed (Participants) | 1
Micrograms per milliliter | 109.59 (NA) — 'NA' indicates that geometric coefficient of variation could not be calculated as only 1 participant was analyzed.

13. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), and AEs of Special Interest (AESIs) Through Week 12
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in the offspring of a study participant; or other situations as per medical and scientific judgement of the Investigator. AESIs defined in the protocol included post-injection systemic reactions and hypersensitivity reactions, infections of special interest, malignancies, and depression, suicidality, or self-injury. Number of participants with AEs, SAEs, and AESIs has been reported.
Time Frame: Up to Week 12
Population: Intent-to-Treat (ITT) Analysis Set included all participants assigned treatment who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg/mL
Number analyzed (Participants) | 16
Participants
  AEs | 13
  SAEs | 0
  AESIs | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs, and non-SAEs were collected up to 28 weeks (treatment: up to 12 weeks and follow-up: up to 16 weeks)
Description: All-cause mortality, SAEs, and non-SAEs were analyzed for ITT Analysis Set that included all participants assigned treatment who received at least one dose of study treatment.
Arm/Group | Belimumab 200 mg/mL
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 13/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab 200 mg/mL (N=16)
Upper respiratory tract infection (Infections and infestations) | 9 (17)
Bronchitis (Infections and infestations) | 3 (3)
Bacterial infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Mycoplasma infection (Infections and infestations) | 1 (1)
Tinea versicolour (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
White blood cell count decreased (Investigations) | 1 (2)
Weight fluctuation (Metabolism and nutrition disorders) | 1 (1)
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT05917288/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT05917288/SAP_001.pdf